CLINICAL TRIAL: NCT03943381
Title: Duplex US in Pelvic Congestion Syndrome in Females
Brief Title: Duplex US in Pelvic Congestion Syndrome in Females (PCS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed AbuDeif Sayed, Dr, Principal Investigator., Assiut University
Other Study IDs: Duplex US in PCS
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Pelvic Pain Syndrome
Keywords: PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Duplex US — Duplex US (Caliper, wave forms...)in evaluation of Pelvic Veins (namely left ovarian vein). in pelvic congestion syndrome

SUMMARY:
To investigate the feasibility of Duplex US in Diagnosis of Pelvic Congestion Syndrome

DETAILED DESCRIPTION:
* In the past, a diagnosis of chronic pelvic pain left many women frustrated with few treatment options and a lack of available resources. Their physicians were likewise perplexed, despite the endless acquisition of negative laboratory and imaging data as well as inconclusive consultations obtained. In the last 10 years, improved scientiﬁc understanding and increased physician awareness have lessened the confusion surrounding this condition and its distinct association with pelvic congestion syndrome (PCS). Furthermore, reﬁnements of medical and minimally invasive surgical solutions give affected patients more therapeutic choices today.
* Since anatomical venous variations in the pelvis are common, it is important to know the anatomy of these vessels for treatment planning. Imaging is critical in the evaluation of pelvic varices, both to differentiate them from other condition and also because pelvic varices may be secondary to serious underlying pathology, such as inferior vena caval obstruction, portal hypertension, increased pelvic blood flow, and vascular malformations.

Sonographic findings of pelvic congestion syndrome were dilated left ovarian vein with reversed caudal flow, presence of varicocele, dilated arcuate veins crossing the uterine myometrium, polycystic changes of the ovary, and variable duplex waveform during the Valsalva's maneuver. Combined transabdominal and transvaginal sonography are potentially useful as a noninvasive screening & grading tool for determining which patients with chronic pelvic pain may benefit from selective ovarian venography and transcatheter embolization

ELIGIBILITY:
Inclusion Criteria:

* All patients with signs and symptoms of PCS

Exclusion Criteria:

* No

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — In the past, a diagnosis of chronic pelvic pain left many women frustrated with few treatment options and a lack of available resources. Their physicians were likewise perplexed, despite the endless acquisition of negative laboratory and imaging data as well as inconclusive consultations obtained. In the last 10 years, improved scientiﬁc understanding and increased physician awareness have lessened the confusion surrounding this condition and its distinct association with pelvic congestion syndrome (PCS). Furthermore, reﬁnements of medical and minimally invasive surgical solutions give affected patients more therapeutic choices today
Study Population: females with chronic lower abdominal pain, signs and symptoms of pelvic congestion syndrome
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-05-10 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Duplex US in Pelvic Congestion Syndrome in females | 6 months
  to investigate the feasibility of Duplex US in diagnosis of Pelvic Congestion Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Hossam M Galal, Study Chair — Assiut University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
to be shared when finished